CLINICAL TRIAL: NCT06308848
Title: Proof-of-Concept Study for a Microbiota-Directed Food in Children With Uncomplicated Severe Acute Malnutrition in Rural Bangladesh
Brief Title: Microbiota Directed Food for Children With Severe Acute Malnutrition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-22077
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Severe Acute Malnutrition
Keywords: Microbiota directed food; SAM; Gut microbiota; Bangladesh
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — milk-derived factor

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (Proof of concept study)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiota Directed Food (MDF) (Experimental): Each participant will receive 12 weeks of MDF supplement. After finishing the intervention phase, he/she will be followed-up for a 12-month period.
  Interventions: Dietary Supplement: Microbiota-Directed Food
- Ready-to-Use Therapeutic Food (RUTF) (Active Comparator): Each participant will receive 12 weeks of RUTF supplement. After finishing the intervention phase, he/she will be followed-up for a 12-month period.
  Interventions: Dietary Supplement: Ready-to-Use Therapeutic Food

INTERVENTIONS:
Dietary Supplement: Microbiota-Directed Food — MDF is a microbiota directed food for malnourished children aged 6 months and above. It is in sachet form. The sachet contains 92 gm of supplements and provides approximately 506 kcal.
  Other Names: MDF
  Arms: Microbiota Directed Food (MDF)
Dietary Supplement: Ready-to-Use Therapeutic Food — RUTF is standard ready-to-use therapeutic food for SAM children aged 6 months and above.
  Other Names: RUTF
  Arms: Ready-to-Use Therapeutic Food (RUTF)

SUMMARY:
Severe acute malnutrition (SAM) refers to a condition characterized by a significant deficit in weight-for-length measurements in children aged 6 to 59 months. It is a crucial public health concern with detrimental effects on child growth, development, and overall well-being. Addressing SAM is crucial to prevent its progression to other childhood morbidity and mortality and to ensure healthy child development. To meet the nutritional requirement of SAM children, icddr,b have come up with a novel intervention named microbiota-directed food (MDF), a ready-to-use therapeutic food. The investigators propose this proof-of-concept trial to establish evidence on the effect of this novel intervention on ponderal growth, microbial and proteomic recovery among the children with SAM in comparison to the standard RUTF.

DETAILED DESCRIPTION:
Burden: As per Global Nutrition report 2021, 45.4 million children under the age of 5 years were reported to be wasted. Asia is a home to more than three-quarters of all these children suffering from wasting. According to Bangladesh Multiple Indicator Cluster Survey 2019 around 10% under 5 children were wasted, while 2.3% suffered from severe form of wasting also known as severe acute malnutrition (SAM). SAM is defined by the World Health Organization (WHO) as weight-for-length Z score (WLZ) of less than -3 and/or presence of bilateral pedal edema and/or a mid-upper arm circumference less than 115 mm.

SAM children are found to be suffering from relative gut microbial immaturity, which is related to their growth faltering. Ready-to-use therapeutic food (RUTF) is a key component of the treatment protocol for SAM children and is widely used throughout the world. Which however is found to be partially effective or ineffective in repairing the gut microbial immaturity present in SAM children. To combat this, affordable therapeutic food formulation is needed that can be used to treat acute malnutrition in children with the potential to restore gut microbial colony related to growth and early childhood development.

Knowledge gap: Researchers at icddr,b in collaboration with Washington University in St. Louis has developed a Microbiota-Directed Complementary Food (MDCF) formulation (based on locally available food ingredients) that has the potential of repairing the gut microbiota of children with malnutrition. Results from a recently conducted study of MDCF on Bangladeshi children suffering from moderate acute malnutrition (MAM) showed that the children who received the food exhibited significantly faster rates of ponderal growth compared to those treated with a standard ready-to-use supplementary food. Early evidence, however, is limited to a small sample of children with MAM. This leaves a paucity of data on the role of microbiota directed food interventions on the nutritional as well as microbial recovery and proteomic improvement in children with SAM.

Relevance: To meet the nutritional requirement of SAM children, researchers have come up with a novel intervention named Microbiota-Directed Food (MDF), a ready-to-use therapeutic food by modifying the original MDCF recipe to meet the nutritional requirement of SAM children as well as to make it align with the existing WHO/UNICEF specifications for a nutritional intervention for treating acute malnutrition. The proposed formulation MDF with a relatively lower calorie content will improve the nutritional status by modulating and improving the gut microbial dysbiosis that is present in SAM children. Therefore, the investigators propose this POC trial to generate evidence on the effect of the novel intervention on the ponderal growth, microbial and proteomic recovery among the children with SAM in comparison to the standard RUTF.

Hypothesis: The locally developed MDF would be proven beneficial in nutritional recovery, repairing gut microbiota and restoring plasma biomarkers of healthy growth when compared to standard RUTF among children suffering from SAM.

Primary Objective:

• To assess the role of MDF in improving the weight-for-length Z score (WLZ) of SAM children

Secondary Objectives:

* To investigate the effect of MDF in repairing the gut microbiota of SAM children
* To monitor the change produced by MDF in rebalancing the body composition of the SAM children towards a more appropriate lean-to-fat mass ratio present in SAM children
* To explore the impact of MDF in restoring plasma biomarkers of healthy growth
* To measure the efficacy of MDF in improving the Weight-for-Age Z-score (WAZ) in children with SAM
* To measure the efficacy of MDF in improving the Length-for-Age Z-score (LAZ) in children with SAM
* To assess the acceptability of the MDF among SAM children
* To measure the intake of the MDF by SAM children

Study design:

This will be a double blinded, parallel-group, simple randomized controlled trial.

Study site:

This study will be conducted among residents of Kurigram district. Kurigram District is situated in Northwest Bangladesh (Rangpur Division).

Randomization:

At enrolment, children will be randomized into one of the two intervention arms using permuted block randomization method to ensure even distribution across the intervention arms over time.

Recruitment, Screening and Consenting:

Census, screening, enrolment of study participants will be done in Kurigram. Initially 6-<24 months old children will be screened by the study health workers through community surveillance by measurement of MUAC (measuring weight and length/height where possible) of the children. Parents of eligible children who meet the inclusion criterion will be approached about enrolment into the study. A trained Field Research Assistant will explain the study in detail, answer any questions from the parent(s), and invite the parent(s) to enroll the child in the study. After acquiring consent from the parents, at the beginning of the study, the child along with his parents will be invited to the study clinic where initial anthropometric assessment (weight, length, MUAC) will be done, and they will be assessed further for eligibility by the study medical personnel regarding any concurrent illness. If found eligible an appetite test will be performed among these children. For the appetite test, standard RUTF will be offered to each child. If a child had a body weight of <4 kg, then she/he will be offered an amount of 11.5 g, 23 g will be offered if body weight is between 4 and 9.9 kg, 46 g if between 10 and 14.9 kg and 69 g for those ≥15 kg. A child will be considered to have passed the appetite test if she/he consume the required amount according to his/her body weight within 45 minutes. If a child passes the appetite test, then he or she will be considered for enrolment into the study. Our rationale behind the use of 45 minutes as the duration for the appetite test was based on previously published articles.

If the child passes the appetite test, our study research assistant will sought additional information from the parents on the demographic characteristics (families' wealth, standard of housing, family structure and parental characteristics etc.), household food insecurity (HFIAS), vaccination status of the children.

Intervention delivery and feeding:

The study design comprises a 3-month period of nutritional intervention and 12-month post-intervention follow-up. The recommended nutrition for the SAM children is about 150-200 Kcal/kg/day including breast feeding. As the care providers will encourage the study children to receive the diet while continuing to receive their usual diet, the investigators therefore have set the target intake to be 175 kcal/kg/day as per national and international guidelines. Every child will be provided an appropriate amount of the therapeutic diet (~500kCal/92g sachet) based on their weight from the day of enrolment. Interventions are iso-caloric.

Both the study interventions will be delivered to the homes of participants by project staff on a weekly basis as sachet versions will be produced by a food manufacturing industry. The mother, or the main caregiver will feed the participant at home. The mother/primary caregiver will be instructed to feed the child directly from the sachet. If the child doesn't feel comfortable consuming directly from sachet, they can also spoon or use properly washed hands to feed the diets to their children until s/he refuses to eat. Children will be considered as refusing further intake if they move their head away from the food, cry, clamp the mouth or clinch the teeth, or become agitated, spit out the food or refuse to swallow. Once the child refuses to take, mothers/caregivers will be counselled to give a pause and then try after some time.

Mother/caregiver will be properly trained to monitor their child for any possible side effects/adverse events (e.g., rash, urticaria due to food allergy or any significant changes in clinical status). And if any side effects/adverse events are observed, they will be advised to contact study team immediately. Additionally, the enrolled children will be monitored and caregivers will also be asked every week by trained Field Research Assistants for any illness/side effects/adverse events (e.g., increases in diarrhoea, flatulence, vomiting, skin rash or urticaria due to food allergy or any significant changes in clinical status). If any side effects/adverse events are observed, then they will receive standard care at the nearest health facility or other higher centre if required.

At each weekly food delivery visit, all used and unused food packets from previous week will be collected for weighing in order to estimate intake during the period. In addition, study personnel will ask mothers/caregivers to rate their child's liking of the supplement on 7-point Hedonic scale. A score of 7, will be ranked as 'like extremely' and the lowest value 1 will be ranked as 'dislike extremely'. Hedonic scale data will be collected one week after the initiation of the intervention.

Morbidity data will be collected weekly during the intervention period and bi-weekly during the first three months of the follow-up period.

The Caregiver Reported Early Development Instruments (CREDI) long form will be evaluated for all the children at enrollment, at the end of intervention and three months after finishing intervention.

Food frequency questionnaires (FFQ) will be completed at enrolment, prior to randomization and monthly during the entire intervention period and during the first three months of the follow-up period and three monthly during the rest of the period in order to assess nutrient intake.

Anthropometry:

Anthropometric assessment will be performed by trained study personnel at enrolment, every two weeks interval during the intervention phase and then monthly for the first three months of the follow up period and then at three monthly for the rest of the period until end of the study.

Body composition analysis:

Bioelectrical Impedance Analysis (BIA) is a method of assessing the body composition by measuring the body fat in relation to lean body mass. BIA will be used to measure total fat and fat free at the beginning, at the end of intervention and three months after completing intervention.

Faecal sample collection:

1-2 gm of faecal material will be collected from each child at enrolment, monthly during the intervention period, at the end of intervention and at 4, 5, 6, 9, 12th month during the follow-up period and the end of study.

Blood sample collection:

2 mL of blood samples will be collected from every SAM child at enrolment and just after the intervention is completed and at the 9th month during follow up period and at the end of the study.

Oral swab collection:

Oral swab samples will be collected by using a commercial kit from each child at enrolment, after the intervention/treatment, and at the end of the follow-up period for measuring microbiota.

Standard care All participants will receive standard care at enrolment and throughout the period of the study, including screening for common illnesses and routine medications, as per the national protocol. Standard treatment for community management of severe acute malnutrition as per national guideline. Treatment for all indicated conditions will be provided as per IMCI guidelines and the national protocol free of charge. All concomitant treatments will be recorded in the appropriate study case report form (CRF).

All caregivers will receive basic nutritional and general health counselling at each visit. Caregivers will be provided with information regarding acute malnutrition as well as the benefits of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The trial will include SAM children of either sex without any medical complication
* Children aged between 6-<24 months and with MUAC <115 mm and/or WLZ <-3

Exclusion Criteria:

* Children are not suffering from SAM.
* Children with bi-pedal oedema.
* Failed to obtain consent for study participation from parents or legal guardian.
* Suffering from any chronic illness(es) or having severe anemia (< 8 g/dl).
* History of using antibiotics in the past seven days.
* Children participating in other food intervention programs.
* Children having known history of soy, peanut or milk protein allergy.
* Children who will not pass appetite test.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in Weight-for-Length Z-score (WLZ) | Baseline to 12 weeks of intervention followed by 12 months of follow-up
  In this study, nutritional status will be assessed through anthropometric measurement at enrolment, every two weeks interval during the intervention phase and then monthly for the first three months of the follow up period and then at three monthly for the rest of the period until end of the study.

SECONDARY OUTCOMES:
Gut microbial community repair | Baseline to 12 weeks of intervention followed by 12 months of follow-up
  Non-diarrheal stool samples will be collected at enrolment, monthly during the intervention period, at the end of intervention and at 4, 5, 6, 9, 12th month during the follow-up period and the end of study from all the participants for assessment of the composition of gut microbiota and features of the microbiome.
  Oral swab samples will be collected by using a commercial kit from each child at enrolment, after the intervention/treatment, and at the end of the follow-up period for measuring microbiota.
Improvement in the levels of plasma protein biomarkers of healthy growth | Baseline to 12 weeks of intervention followed by 12 months of follow-up
  Blood samples will be collected at enrolment and just after the intervention is completed and at the 9th month during follow up period and at the end of the study.
  Non-diarrheal stool samples will be collected at enrolment, monthly during the intervention period, at the end of intervention and at 4, 5, 6, 9, 12th month during the follow-up period and the end of study from all the participants for measuring biomarkers of gut inflammation.
Mean change in Weight-for-Age Z-score (WAZ) | Baseline to 12 weeks of intervention followed by 12 months of follow-up
  In this study, nutritional status will be assessed through anthropometric measurement at enrolment, every two weeks interval during the intervention phase and then monthly for the first three months of the follow up period and then at three monthly for the rest of the period until end of the study.
Mean change in Length-for-Age Z-score (LAZ) | Baseline to 12 weeks of intervention followed by 12 months of follow-up
  In this study, nutritional status will be assessed through anthropometric measurement at enrolment, every two weeks interval during the intervention phase and then monthly for the first three months of the follow up period and then at three monthly for the rest of the period until end of the study.
Mean change in body composition (% body fat mass and % fat-free mass) | Baseline to 12 weeks of intervention followed by 3 months of follow-up
  In this study, nutritional status will be also assessed through Bioelectrical impedance at the beginning, at the end of intervention and three months after completing intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Md Hasan Hafizur Rahman, MPH, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Kurigram Study site, Kurigrām, Bangladesh

IPD SHARING:
Plan to Share IPD: No